CLINICAL TRIAL: NCT05942703
Title: Non-interventional Study Exploring the Relationship Between Porphyromonas Gingivalis and Obesity in Patients With Periodontitis
Brief Title: Relationship Between Porphyromonas Gingivalis and Obesity in Patients With Periodontitis
Acronym: PAROBIOTA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/20/0478
Record Dates: First submitted 2022-12-05; First posted 2023-07-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- obese patients: Patients with a body mass index superior or equal at 30 and with a periodontitis
  Interventions: Other: saliva samples
- non-obese (BMI<30) patients: Patients with a body mass index inferior at 30 with a periodontitis
  Interventions: Other: saliva samples

INTERVENTIONS:
Other: saliva samples — Saliva samples, which are part of the usual treatment, will be carried out before and after the non-surgical periodontal treatment
  Other Names: periodontal plaque samples

SUMMARY:
Obesity is recognized as a major public health problem. Recent research suggests the involvement of the gut microbiota in the development of obesity. Indeed, obese people are characterized by a dysbiotic intestinal microbiota. Periodontitis are chronic inflammatory oral pathologies linked to an imbalance between the bacterial etiological factor, oral dysbiosis, and the host's immune defenses.They lead to the destruction of the supporting tissues of the tooth and an apical migration of the periodontal attachment system, thus leading to the formation of the pathognomonic entity of the disease, the periodontal pocket.the presence of bacteria of oral origin such as Porphyromonas gingivalis (Pg) has been demonstrated in the adipose tissue of obese patients inducing a chronic low-grade inflammatory response by macrophages which leads to the proliferation of adipocyte precursors predisposing to obesity. The main objective is to assess the average amount of Porphyromonas gingivalis (Pg) in the saliva of obese people (BMI ≥ 30) with periodontitis.

DETAILED DESCRIPTION:
Obesity is recognized as a major public health problem. Recent research suggests the involvement of the gut microbiota in the development of obesity. Indeed, obese people are characterized by a dysbiotic intestinal microbiota. Periodontitis are chronic inflammatory oral pathologies linked to an imbalance between the bacterial etiological factor, oral dysbiosis, and the host's immune defenses.They lead to the destruction of the supporting tissues of the tooth and an apical migration of the periodontal attachment system, thus leading to the formation of the pathognomonic entity of the disease, the periodontal pocket.the presence of bacteria of oral origin such as Porphyromonas gingivalis (Pg) has been demonstrated in the adipose tissue of obese patients inducing a chronic low-grade inflammatory response by macrophages which leads to the proliferation of adipocyte precursors predisposing to obesity. The main objective is to assess the average amount of Porphyromonas gingivalis (Pg) in the saliva of obese people (BMI ≥ 30) with periodontitis.This study is a comparative cross-sectional non-interventional study with retrospective and prospective and consecutive recruitment of participants.

Prospective patient recruitment:

During the patient's visit to the periodontology department, if the patient has periodontitis and has given his non-objection, he will be included in the study. A routine check-up in odontology will then be carried out: complete medical questionnaire (general, hygiene and dietetics), clinical examination (visual examination and statement of periodontal indices), radiological examination. Samples of saliva and periodontal plaque, conventionally taken in current dental surgery practice in the periodontal management of patients, will be used to carry out bacterial assays. CThe saliva samples, which are part of the usual treatment, will be carried out before and after the non-surgical periodontal treatment.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old
* having periodontitis
* able to receive information on the course of the study and to understand the information form to participate in the study.
* having given their non-objection to participate in the study

Exclusion Criteria:

* Having taken antibiotics, prebiotics or probiotics in the month prior to inclusion
* During pregnancy or breastfeeding
* With a history of oral surgery in the month prior to inclusion
* At risk of infection (existence of one or more known chronic infectious diseases)
* Suffering from a general pathology contraindicating the performance of diagnostic procedures such as periodontal probing (patients at high risk of infective endocarditis according to the French National Agency for the Safety of Medicines and Products of Health ANSM)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: any patient coming for consultation in the periodontology department
Sampling Method: Non-Probability Sample
Enrollment: 311 (Estimated)
Dates: Start 2022-12-05 (Actual); Primary Completion 2024-03-27 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Analysis by bacterial culture and taxonomic analysis (MiSEQ) of the microbiological composition of saliva | 8 weeks
  Assess the microbiological composition of saliva and periodontal plaque in obese (BMI≥30) and non-obese (BMI<30) patients with periodontitis.
Analysis by bacterial culture and taxonomic analysis (MiSEQ) of the microbiological composition periodontal plaque | 8 weeks
  Assess the microbiological composition of periodontal plaque in obese (BMI≥30) and non-obese (BMI<30) patients with periodontitis.

CONTACTS AND LOCATIONS:
Overall Officials: Sara LAURENCIN, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- UHToulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No